CLINICAL TRIAL: NCT05862558
Title: Intravascular Lithotripsy in High Risk Calcified Iliac Anatomy for Transfemoral TAVR
Acronym: ILIT
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 022-277
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Iliac Disease; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Shockwave Balloon — Intravascular lithotripsy (IVL) performed with the Shockwave balloon (Shockwave Medical Inc) enables treatment of calcified stenosis of the peripheral arteries by using sonic pressure waves to selectively disrupt superficial and deep calcium without impacting healthy tissue

SUMMARY:
To assess the efficacy and safety of Intravascular Lithotripsy (IVL) in subjects undergoing transfemoral TAVR in patients with severe iliac disease, prohibitive for transfemoral TAVR in patients with severe symptomatic aortic stenosis, otherwise considered for alternative access TAVR. (e.g. trans-carotid)

DETAILED DESCRIPTION:
The goal of this post-market, prospective, observational single-arm cohort study is to assess the efficacy and safety of Intravascular Lithotripsy (IVL) in subjects undergoing transfemoral TAVR in patients with severe iliac disease, prohibitive for transfemoral TAVR in patients with severe symptomatic aortic stenosis, otherwise considered for alternative access TAVR. (e.g. trans-carotid). This is a study of patients referred to BSW The Heart Hospital, Plano for evaluation of critical aortic stenosis. Those planned to undergo TAVR, have prohibitive iliofemoral disease, and otherwise considered for alternative access, will be considered for the study. The medical devices being used are in the post-market stage as it is being used in accordance with its approved labeling, treating iliofemoral disease.

Study data will be recorded prospectively on dedicated Data Collection Forms and stored locally in a secure format. De-identified data will be uploaded for statistical analysis. IRB approval for the study will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 90 years of age, inclusive, at the time of signing the informed consent
2. Iliofemoral disease warrants treatment, per routine guidelines (greater than 50% stenosis and heavy calcification of the iliac's).
3. Severe symptomatic aortic stenosis and undergoing a planned TAVR procedure
4. Prohibitive iliofemoral disease, as determined by the diagnostic CT abdomen and pelvis.
5. Subjects can provide written, informed consent.

Exclusion Criteria:

1. Subject is participating in another research study involving an investigational agent that has not reached the primary endpoint.
2. Subject who has contraindications to IVL
3. Subject who has contraindications or is not eligible for TAVR

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must meet the inclusion criteria and have none of the exclusion criteria to be eligible for participation in this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Acute technical success per the DISRUPT PAD definition at the time of intervention | At time of IVL procedure
  Defined as final residual stenosis ≤30% without flow-limiting dissection (≥ Grade D) of the lesion
Success rate of transfemoral delivery of a TAVR system post IVL within 30 days of treatment | At the time of TAVR procedure
  To know the efficacy of the treatment

SECONDARY OUTCOMES:
Applicable VARC-3 criteria at the time of peripheral intervention for bleeding, access site and access related complications. | At IVL procedure
  To understand the efficacy of the treatment
Major adverse events within 1 year | 1 year after IVL procedure
  need for emergency surgical revascularization of target limb, unplanned target limb major amputation (above the ankle), symptomatic thrombus or distal emboli that requires surgical, mechanical, or pharmacologic means to improve flow and extend hospitalization, perforations that require an intervention, including bail-out stenting.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott and White Heart Hospital, Plano, Texas, United States

REFERENCES:
- [Result] Junquera L, Kalavrouziotis D, Cote M, Dumont E, Paradis JM, DeLarochelliere R, Rodes-Cabau J, Mohammadi S. Results of transcarotid compared with transfemoral transcatheter aortic valve replacement. J Thorac Cardiovasc Surg. 2022 Jan;163(1):69-77. doi: 10.1016/j.jtcvs.2020.03.091. Epub 2020 Apr 13. PMID 32387164
- [Result] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Result] Ristalli F, Dini CS, Stolcova M, Nardi G, Valente S, Meucci F, Di Mario C. Role of Lithotripsy for Small Calcified Iliacs in the Era of Big Devices. Curr Cardiol Rep. 2019 Nov 22;21(11):143. doi: 10.1007/s11886-019-1245-2. PMID 31758362
- [Result] Kumar N, Khera R, Fonarow GC, Bhatt DL. Comparison of Outcomes of Transfemoral Versus Transapical Approach for Transcatheter Aortic Valve Implantation. Am J Cardiol. 2018 Nov 1;122(9):1520-1526. doi: 10.1016/j.amjcard.2018.07.025. Epub 2018 Aug 7. PMID 30190074
- [Result] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Munoz DR, Rosenhek R, Sjogren J, Mas PT, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL. 2017 ESC/EACTS Guidelines for the Management of Valvular Heart Disease. Rev Esp Cardiol (Engl Ed). 2018 Feb;71(2):110. doi: 10.1016/j.rec.2017.12.013. No abstract available. English, Spanish. PMID 29425605
- [Result] Rogers T, Gai J, Torguson R, Okubagzi PG, Shults C, Ben-Dor I, Satler LF, Waksman R. Predicted magnitude of alternate access in the contemporary transcatheter aortic valve replacement era. Catheter Cardiovasc Interv. 2018 Nov 1;92(5):964-971. doi: 10.1002/ccd.27668. Epub 2018 Jul 18. PMID 30019839
- [Result] Di Mario C, Goodwin M, Ristalli F, Ravani M, Meucci F, Stolcova M, Sardella G, Salvi N, Bedogni F, Berti S, Babaliaros VC, Pop A, Caparrelli D, Stewart J, Devireddy C. A Prospective Registry of Intravascular Lithotripsy-Enabled Vascular Access for Transfemoral Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2019 Mar 11;12(5):502-504. doi: 10.1016/j.jcin.2019.01.211. No abstract available. PMID 30846091
- [Result] Kassimis G, Didagelos M, De Maria GL, Kontogiannis N, Karamasis GV, Katsikis A, Sularz A, Karvounis H, Kanonidis I, Krokidis M, Ziakas A, Banning AP. Shockwave Intravascular Lithotripsy for the Treatment of Severe Vascular Calcification. Angiology. 2020 Sep;71(8):677-688. doi: 10.1177/0003319720932455. Epub 2020 Jun 22. PMID 32567327
- [Result] Cruz-Gonzalez I, Gonzalez Ferreiro R, Martin Moreiras J, Trejo Velasco B, Barreiro Perez M, Diego Nieto A, Herrero Garibi J, Rodriguez Collado J, Sanchez Fernandez PL. Facilitated Transfemoral Access by Shockwave Lithoplasty for Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2019 Mar 11;12(5):e35-e38. doi: 10.1016/j.jcin.2018.11.041. Epub 2019 Feb 13. No abstract available. PMID 30772295
- [Result] Gorla R, Cannone GS, Bedogni F, De Marco F. Transfemoral aortic valve implantation following lithoplasty of iliac artery in a patient with poor vascular access. Catheter Cardiovasc Interv. 2019 Feb 15;93(3):E140-E142. doi: 10.1002/ccd.27812. Epub 2018 Sep 9. PMID 30196575
- [Result] Sawaya FJ, Bajoras V, Vanhaverbeke M, Wang C, Bieliauskas G, Sondergaard L, De Backer O. Intravascular Lithotripsy-Assisted Transfemoral TAVI: The Copenhagen Experience and Literature Review. Front Cardiovasc Med. 2021 Sep 22;8:739750. doi: 10.3389/fcvm.2021.739750. eCollection 2021. PMID 34631837
- [Result] Price LZ, Safir SR, Faries PL, McKinsey JF, Tang GHL, Tadros RO. Shockwave lithotripsy facilitates large-bore vascular access through calcified arteries. J Vasc Surg Cases Innov Tech. 2020 Sep 12;7(1):164-170. doi: 10.1016/j.jvscit.2020.09.002. eCollection 2021 Mar. PMID 33748555